CLINICAL TRIAL: NCT02729558
Title: Postoperative Local Stereotactic Radiotherapy Versus Observation Following a Complete Resection of a Single Brain Metastasis
Brief Title: Local Radiotherapy Following Complete Resection of a Brain Metastasis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Too limited accrual
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: The Netherlands Cancer Institute (Other); UMC Utrecht (Other)
Responsible Party: Principal Investigator, Anna Bruynzeel, MD PhD Radiation Oncologist, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL5128302914
Record Dates: First submitted 2016-02-19; First posted 2016-04-06 (Estimated); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Brain Neoplasms
Keywords: brain metastases; radiotherapy; resection
MeSH Terms: conditions — Brain Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- observation (No Intervention): Watchful waiting
- local stereotactic radiotherapy (SRT) (Active Comparator): local SRT in three fractions of 8 Gy to the surgical cavity
  Interventions: Radiation: local SRT

INTERVENTIONS:
Radiation: local SRT — local stereotactic radiotherapy in three fractions of 8 Gy to the surgical cavity
  Other Names: stereotactic radiotherapy; radiosurgery
  Arms: local stereotactic radiotherapy (SRT)

SUMMARY:
Objective: To improve local control following complete resection of a single brain metastasis using fractionated local stereotactic radiotherapy, whilst maintaining neurological functioning, neurocognition and quality of life.

Study design: Multicenter randomized phase III, with at least three high-volume Dutch centers participating in the trial. Stratification on primary tumor type and age.

Study population: Patients undergoing complete resection of a single brain metastasis, confirmed by an early (i.e. within 72 hours) postoperative contrast-enhanced MR scan.

Study intervention: Patients will be randomized between observation alone (standard arm) and local stereotactic radiotherapy in three fractions of 8 Gy to the surgical cavity (study arm).

Main study parameters: Primary objective: local control rate at 6 months. Secondary objectives: local control rate at 12 months, neurological functioning, freedom from clinical neurological progression, performance status, quality of life, toxicity, steroid use, neurocognition and overall survival.

DETAILED DESCRIPTION:
The objective of this study is to improve local control following complete resection of a single brain metastasis of solid tumors using fractionated local stereotactic radiotherapy, whilst maintaining neurological functioning, neurocognition and quality of life. The study is performed in the form of a multicenter randomized phase III, with at least three high-volume Dutch centers participating in the trial. Stratification will be performed on primary tumor type and age. A total of 70 patients will be included. Inclusion is restricted to patients who underwent a complete resection of a single brain metastasis, confirmed by an early (i.e. within 72 hours) postoperative contrast-enhanced magnetic resonance (MR) scan. Patients will be randomized between observation alone (standard arm) and local stereotactic radiotherapy in three fractions of 8 Gy to the surgical cavity (study arm).The main study parameters are: local control rate at 6 months (primary outcome measure) and local control rate at 12 months, neurological functioning, freedom from clinical neurological progression, performance status, quality of life, toxicity, steroid use, neurocognition and overall survival (secondary outcome measures). Follow up will be performed at three-monthly interval during the first two years, including MRI scans. Quality of life questionaires and neurocognitive functioning tests will be performed at fixed intervals during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older.
* Radiologically confirmed complete resection of a single brain metastasis on a contrast-enhanced MRI within 72 h after resection.
* Primary solid tumor, excluding hematologic malignancy, germ cell tumor, small cell lung cancer.
* Stable extracranial tumor (primary tumor and/or systemic metastases) during the last three months with or without treatment or progressive extracranial tumor and/or systemic metastases for which effective treatment is available.
* World Health Organization (WHO) performance score 0-2.
* Ability to provide written informed consent.

Exclusion Criteria:

* Prior treatment for brain metastases (i.e. surgery, stereotactic radiotherapy or WBRT).
* Distant brain metastases or radiological findings on MRI suspected for leptomeningeal tumor spread on the postoperative MRI.
* Concurrent use of systemic therapy during local stereotactic radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
local control rate | at 6 months
  as assessed on follow-up MRI scans

SECONDARY OUTCOMES:
Decrease in neurocognitive test results using the Hopkins Verbal Learning Test Revised (HVLT-R), in full cohorts | baseline, at 3 months, 6 months and 12 months
  Neurocognitive testing will be performed at baseline, at three, six and twelve months follow-up using the Hopkins Verbal Learning Test Revised (HVLT-R). The HVLT-R is one of the components used to form the core set of cognitive tests recommended to use in oncology trials. This test measures immediate memory span, provides a learning curve, measures both short-term and longer-term retention, and allows for a comparison between retrieval efficiency and learning. This version includes 3 learning trials of a 12-word list, an interval of 20 minutes a delayed recall, and a recognition trial consisting of the target words interspersed with distractor words. The score on the recognition trial is the total number of correct response. This measure has adequate psychometric properties and 6 multiple forms.
Decrease in specified neurocognitive test results using the Trail Making A and B, in full cohorts | baseline, at 3 months, 6 months and 12 months
  Neurocognitive testing will be performed at baseline, at three, six and twelve months follow-up using the Trail Making A and B. This test is one of the components used to form the core set of cognitive tests recommended to use in oncology trials. This is a test of visual conceptual and visuomotor tracking. It measures psychomotor speed and aspects of executive function. It is given in two parts, A and B. The subject must first draw lines to connect consecutively numbered circles on one work sheet (part A) and then connect the same number of consecutively numbered and lettered circles on another worksheet by alternating between the two sequences (part B). The subject is urged to connect the circles as fast as possible
Decrease in neurocognitive test results using the Controlled Oral Word Association (COWA), in full cohorts | baseline, at 3 months, 6 months and 12 months
  Neurocognitive testing will be performed at baseline, at three, six and twelve months follow-up using the Controlled Oral Word Association (COWA). The COWA is one of the components used to form the core set of cognitive tests recommended to use in oncology trials. This test measures speeded verbal fluency and aspects of executive function. In this test, subjects are asked to generate as many words as possible in 1 minute beginning with "B", "D," and "H". It has two forms.
Decrease in neurocognitive test results using using the Wechsler Adult Intelligence Scale (WAIS) III Digit Span and WAIS III Digit Symbol, in full cohorts | baseline, at 3 months, 6 months and 12 months
  Neurocognitive testing will be performed at baseline, at three, six and twelve months follow-up using the WAIS III Digit Span and WAIS III Digit Symbol. These added cognitive tests are also chosen based on their proven sensitivity to measure change in neuro-oncology patients. The subtest of the WAIS-III (Digit Span) involves forward and backward repetitions of series of digits and provides measures of concentration. This measure has adequate psychometric properties.
  The subtest of the WAIS III (Digit Symbol) involves a symbol substitution task that requires visual-motor coordination, motor persistence, and sustained attention. The test is used as a test for information processing speed. The task consists of pairing numbers to nonsense symbols as quickly as possible.
Decrease in neurocognitive test results using the Grooved Pegboard, in full cohorts | baseline, at 3 months, 6 months and 12 months
  Neurocognitive testing will be performed at baseline, at three, six and twelve months follow-up using the Grooved Pegboard. This added cognitive test is also chosen based on its proven sensitivity to measure change in neuro-oncology patients. This test measures motor speed and dexterity and is an adjusted version of the Purdue Pegboard test. The test consists out of plywood with 2 columns of 30 holes and a zinced bowl filled with metal pegs above each column. Subjects are offered one minute to put as many pegs as possible into the holes. The test has two different trials: dominant hand only and non-dominant hand only.

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Netherlands Cancer Institute - Antoni van Leeuwenhoek, Amsterdam
  - VU University medical center, Amsterdam

IPD SHARING:
Plan to Share IPD: No